CLINICAL TRIAL: NCT04973995
Title: Research on Optimization of Rotator Cuff Injury Diagnosis Plan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021099
Record Dates: First submitted 2021-07-21; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Rotator Cuff Injury
Keywords: physical examination; Rotator cuff; LHBT
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Patients with shoulder pain who received ER lag sign
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received External rotation resistence strength test
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received Patte's test
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received Errsair test
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received speed test
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received Yergason test
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received backward traction test
  Interventions: Behavioral: several physical examinations
- Patients with shoulder pain who received Cui's test
  Interventions: Behavioral: several physical examinations

INTERVENTIONS:
Behavioral: several physical examinations — By using physical examinations, the incidence of these physical examinations corresponding to shoulder muscls injury

SUMMARY:
Rotator cuff injury is a common cause of shoulder pain and dysfunction. Finding out patients with suspected rotator cuff injuries through physical examination of the shoulder joints, MRI further assists in the diagnosis, and final surgical diagnosis and treatment are the current standardized procedures.

How to apply multiple physical examination programs to make judgments sensitively, efficiently and accurately is a clinical problem that needs to be solved urgently.

DETAILED DESCRIPTION:
Rotator cuff injury is a common cause of shoulder pain and dysfunction. The common symptoms of rotator cuff injury include shoulder pain, weakness, and limited mobility. Arthroscopic exploration is the gold standard for the diagnosis of rotator cuff injury, but it is an invasive examination that is difficult to carry out routinely; MRI is sensitive in diagnosing rotator cuff tears Both sex and specificity are high, but due to the popularity, cost and waiting time, it is difficult to be used as a routine screening method.

Therefore, finding patients with suspected rotator cuff injuries through physical examination of the shoulder joints, MRI further assisting in the diagnosis, and final surgical diagnosis and treatment are the current standardized procedures.

However, although there are many physical examination methods for the shoulder joint, the accuracy of each method is different, and each has its own sensitivity and specificity. How to apply multiple examination programs in combination to make it sensitive, efficient and accurate Judgment is a problem that needs to be solved clinically.

This study is expected to adopt prospective research methods to collect and collect patient medical records, preoperative physical examination results, imaging data, and findings during intraoperative exploration, to understand the impact of various shoulder joint physical examination methods and imaging data on rotator cuff injuries

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prepared to undergo arthroscopic surgery for shoulder injuries

Exclusion Criteria:

* Shoulder stiffness, shoulder instability, calcified tendinitis, past surgery, side-to-shoulder disease, hamada osteoarthritis, frozen shoulder, acute joint injury, rheumatoid arthritis, hyperuricemia

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with shoulder pain who were treated at peking university's Third Hospital outpatient clinic for a continuous period of time
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
the Accuracy of different physical examinations | 1week
  After apply these physical examinations, by using Arthroscopic examination find the accuracy of these physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, MD, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No